CLINICAL TRIAL: NCT06166849
Title: Clinical Study of Tooth Enamel Remineralization Using DoReMin Product
Brief Title: Clinical Evaluation of an Experimental Remineralization Product
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL4182693
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: White Spot Lesion
Keywords: white spot lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Fluoride Application (Experimental): Two-step system, consisting of Component A (ammonium fluoride solution) and Component B (calcium fluoride application)
  Interventions: Device: Experimental Fluoride Application
- No Treatment (No Intervention)

INTERVENTIONS:
Device: Experimental Fluoride Application — The two-step system, consisting of Component A and Component B, will be applied once on the white spot lesions
  Arms: Experimental Fluoride Application

SUMMARY:
The study is designed as a split-mouth randomised controlled study. This means within the mouth of one patient one tooth with an initial lesion is treated and coated with the Experimental Remineralization product whereas another comparable tooth with an initial lesion is left untreated. Patients are included upon meeting the inclusion criteria as defined for this clinical trial. In the test group, a remineralization of the incipient carious lesion is expected. The patients are recalled after 1 day (optional), 4 weeks, 4 months and finally after 1 year to evaluate the untreated and treated lesion.

ELIGIBILITY:
Inclusion Criteria:

* At least two incipient carious lesions on the buccal or oral surface of a permanent tooth. Neighbouring teeth should not be in two different groups. There is no maximum amount of lesions.
* Active caries lesion
* Patient at risk of caries
* Vital teeth

Exclusion Criteria:

* Pregnancy
* Enamel detachment at the site of investigation
* Allergies (DoReMin)
* Chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
White Spot Measurement | Baseline to 1 Year
  Analysis of incipient caries or demineralized enamel by using laser fluorescence technology.
ICDAS II visual scoring system (Codes) | Baseline to 1 Year
  Evaluation of the clinical status of the lesions:
  0: Sound tooth surface: No evidence of caries after 5 sec air drying
  1. First visual change in enamel: Opacity or discoloration (white or brown) is visible at the entrance to the pit or fissure seen after prolonged air drying
  2. Distinct visual change in enamel visible when wet, lesion must be visible when dry
  3. Localized enamel breakdown (without clinical visual signs of dentinal involvement) seen when wet and after prolonged drying
  4. Underlying dark shadow from dentin
  5. Distinct cavity with visible dentin
  6. Extensive (more than half the surface) distinct cavity with visible dentin

CONTACTS AND LOCATIONS:
Overall Officials: Ada Delean, Prof. Dr., Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy
Locations (1):
- Iuliu Hatieganu, University of Medicine and Pharmacy, Cluj-Napoca, Romania